CLINICAL TRIAL: NCT01041339
Title: ST Elevation (Acute Coronary Syndrome Versus Pericarditis;Could Measurement of Lp-associated PLA2 -a Vascular Specific Marker of Inflammation- be Helpful to the Clinician?
Brief Title: ST Elevation in Acute Chest Pain; Could Measurement of Lipoprotein-associated Phospholipase A2 (Lp-PLA2) be Helpful to the Clinician?
Status: Completed | Type: Observational
Sponsor: Alexhander Izhaki (Other Government)
Responsible Party: Sponsor-Investigator, Alexhander Izhaki, MD, Wolfson Medical Center
Organization: Wolfson Medical Center (Other Government)
Other Study IDs: 0075-09-WOMC
Record Dates: First submitted 2009-12-30; First posted 2009-12-31 (Estimated); Last update posted 2015-12-15 (Estimated); Status verified 2011-06

CONDITIONS: Acute Chest Syndrome
Keywords: LpPLA2; ST elevation; acute pericarditis
MeSH Terms: conditions — Acute Chest Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma kept in -80 celsius refrigerator
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- acute chest pain ST elevation: patients admitted with acute chest pain sharing ST elevation in ER-ECG and elevated troponin
- controls: asymptomatic patients

SUMMARY:
A blood test (2-3 cc peripheral venous blood) drawn /used from already available required lab tests to distinguish between pericarditis accompanied with electrocardiogram (ECG) signs mimicking infarction. A test of clinical potential if proven to be able to support either origin of acute chest pain etiology.

DETAILED DESCRIPTION:
Too many times young patients presenting with acute chest pain are referred to invasive angiography or treated with anticoagulation therapy a measure of detrimental effect in those inflicted with acute pericarditis.

A simple blood test (the PLAC test) may have some value in aiding rapid diagnosis saving need for cath.

ELIGIBILITY:
Inclusion Criteria:

* acute chest pain
* acute ST elevation
* elevated troponin I

Exclusion Criteria:

* patients with recent (> 24 hour chest pain) myocardial infarction
* refusing to provide blood samples

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: acute chest pain patients admitted to ICCU with acute ST elevation and elevated troponin
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2010-01; Primary Completion 2011-11 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander J Izhaki, MD, Principal Investigator — The E.Wolfson MC
Locations (1):
- The E.Wolfson MC, Holon, Israel

REFERENCES:
- See also: Mayo Clin Proc. 2009;84(1):11-5. — http://www.ncbi.nlm.nih.gov/pubmed/19121248?itool=EntrezSystem2.PEntrez.Pubmed.Pubmed_ResultsPanel.Pubmed_RVDocSum&ordinalpos=1